CLINICAL TRIAL: NCT02595190
Title: A Randomized Controlled Trial to Compare the Efficacy of Medicine Conservative Treatment and Surgical Treatment for Symptomatic Sacral Perineurial Cysts (Tarlov Cysts) and the Applied Value of Resting State Functional Magnetic Resonance Imaging (rfMRI).
Brief Title: Treatment of the Symptomatic Sacral Perineurial Cysts
Acronym: TSSPC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Jiangkai Lin, Vice chief of Neurosurgery Department, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: No.29SROSWH-2015
Record Dates: First submitted 2015-10-23; First posted 2015-11-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Pain
Keywords: Sacral perineurial cysts(Tarlov Cysts); Resting state functional magnetic resonance imaging (rfMRI); VAS; Medicine conservative treatment; Surgical treatment
MeSH Terms: conditions — Pain | interventions — Gabapentin; Tramadol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- surgery group (Experimental): sacral canal cyst microscopic tamponade treatment; resting state functional magnetic resonance imaging (rfMRI)
  Interventions: Procedure: sacral canal cyst microscopic tamponade; Device: resting state functional magnetic resonance imaging (rfMRI)
- drug group (Experimental): gabapentin + tramadol tablets; resting state functional magnetic resonance imaging (rfMRI)
  Interventions: Drug: gabapentin + tramadol; Device: resting state functional magnetic resonance imaging (rfMRI)
- control group (Placebo Comparator): resting state functional magnetic resonance imaging (rfMRI)
  Interventions: Device: resting state functional magnetic resonance imaging (rfMRI)

INTERVENTIONS:
Procedure: sacral canal cyst microscopic tamponade — sacral canal cyst microscopic tamponade treatment
  Arms: surgery group
Drug: gabapentin + tramadol — dose range：gabapentin 400-1200mg tid, tramadol 100-200mg bid
  Arms: drug group
Device: resting state functional magnetic resonance imaging (rfMRI) — First time:2 days before Surgery or Drug use; Second time:3 months after Surgery or Drug use; Third time:1 year after Surgery or Drug use

SUMMARY:
There are very few data and analysis in the literature regarding the symptomatic sacral perineurial cysts. Most studies are case reports or small retrospective sample, which rarely more than 20 cases. There is no an consensus on the choice of treatment (medicine conservative treatment and surgical treatment) for symptomatic sacral perineurial cysts.Our aim, therefore, is to compare the efficacy of medicine conservative treatment and surgical treatment for symptomatic sacral perineurial cysts by a randomized controlled trial. Meanwhile, resting-state functional magnetic resonance imaging is used to detect the changes at pain related brain areas, which will be develop an objective method to evaluate the clinical curative effect of the two treatment options.

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosed with symptomatic sacral perineurial cysts(e.g., lumbosacral or perineal pain, fecal or urinary functions change, sexual function change, lower limb radiation pain, muscle abate, paresthesia, etc)
* 2. Visual analog scale more than or equal to 4
* 3. Signed the informed consent
* 4. Years, range 18-60
* 5. Self-rating anxiety scale (SAS) and self-rating depression scale (SDS) scores < 50
* 6. No Congenital,Mental and other Nervous system diseases
* 7. No Serious Cardiac,Pulmonary,Hepatic and Nephritic disease
* 8. No history of drug allergy
* 9. No pain(including dysmenorrhea) or drug use (e.g., antipyretics,sleeping pills) within the last month
* 10. MRI finding of sacral perineurial cysts, but without any clinical symptoms, included in the negative control group
* 11. MRI finding healthy volunteers don't have sacral perineurial cysts, included in the negative control groupblank control group

Exclusion Criteria:

* 1. Patients with lumbar common diseases(e.g., Lumbar disc, Lumbar spinal stenosis, Lumbar slippage, etc)
* 2. Researchers think that Patients with disease may be interference results(e.g., Spinal deformity, spine fracture, ankylosing spondylitis, spinal tuberculosis and spinal infection, spinal tumor, pelvic inflammatory disease and other disease of department of gynaecology, etc)
* 3. Patients with other nervous system diseases(e.g., cerebral tumor, neurinoma, trigeminal neuralgia,etc)
* 4. Patients with Magnetic resonance imaging contraindication ,including claustrophobic syndrome patients
* 5. Patients with recent (less than 3 years) use chemical drugs or have obvious psychological problems
* 6. In the past 2 months involved in other drugs or devices clinical trials

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2015-03; Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale(VAS) | 3year
Structure and Function connection change(e.g., increase or decrease the thickness of the cortex, or gray matter;function connection increase or decrease) at somatosensory area | 1year

SECONDARY OUTCOMES:
Modify Japanese orthopedic association low back pain score (M-JOA) | 3year
Oswestry Disability Index score (DOI) | 3year
MacNab curative effect evaluation | 3year

OTHER OUTCOMES:
Size of the cyst | 3year
Number of the cyst | 3year
Urine dynamics change(e.g., urinary flow rate) | 3year
Perianal electromyography change | 3year

CONTACTS AND LOCATIONS:
Overall Officials: jiangkai lin, PhD, Principal Investigator — Neurosurgery department of Southwest Hospital,China
Locations (1):
- Southwest Hospital, Chongqing, China